CLINICAL TRIAL: NCT00152464
Title: The Early Prevention of Asthma in Atopic Children (EPAAC™) Study. A Multi-country, Double Blind, Placebo (PLC) Controlled, Randomized, Parallel Group Trial: Evaluation of the Efficacy and Safety of Levocetirizine (LCTZ) (5 mg/ml Oral Drops -0.125 mg/kg b.w. b.i.d.) Administered for 18 Months in Preventing the Onset of Asthma in 12 to 24 Months Old Children Who Suffer From Atopic Dermatitis and Are Sensitized to Grass Pollen and / or House Dust Mite Allergens.
Brief Title: Prevention of Asthma With Levocetirizine 18 Month Treatment in Infants (12 - 24 Months) Suffering From Eczema (Atopic Dermatitis) and Sensitized to Grass Pollen and/or House Dust Mite (HDM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A00309
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Dermatitis, Atopic
Keywords: EPAAC; Atopic children; Asthma; XYZAL; Levocetirizine
MeSH Terms: conditions — Dermatitis, Atopic; Asthma | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levocetirizine (LCTZ) (Experimental): 0.125 mg/kg of Levocetirizine (LCTZ) were administered as oral drops twice daily.
  Interventions: Drug: Levocetirizine
- Placebo (PBO) (Placebo Comparator): Placebo was administered as oral drops twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Pharmaceutical form: Oral drops Route of administration: Oral use
  Arms: Placebo (PBO)
Drug: Levocetirizine — Pharmaceutical form: Oral drops Concentration: 5 mg/ml Route of administration: Oral use
  Other Names: Xyzal
  Arms: Levocetirizine (LCTZ)

SUMMARY:
The Early Prevention of Asthma in Atopic Children (EPAAC™). 24 months study to evaluate the efficacy and safety of levocetirizine (LCTZ) in preventing the onset of asthma in 12 to 24 months old children.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria which must be verified during screening visit (V1):

* Children of either sex aged between 12 and 24 months
* Subjects suffering from symptoms of Atopic Dermatitis (AD) lasting cumulatively for at least 2 months since birth
* Modified Severity Scoring of Atopic Dermatitis (SCORAD) Index >= 10
* Subjects whose biological mother or father, or one sibling has a well-documented history of atopy (AD, allergic rhinitis or asthma)

Inclusion criteria which must be verified during randomization (V2):

* Results of the Radio-allergosorbant (RAST) test for grass pollen (GP) and house dust mite (HDM) are available and Immunoglobulin E (IgE) level against GP >= 0.35 kUA/l and/or IgE level against HDM ≥ 0.35 kUA/l
* Safety laboratory results are within the normal range of the central laboratory or considered as not clinically significant or study disease related by the Investigator

Exclusion Criteria:

Exclusion criteria to verify at screening visit (V1):

Are to be excluded from the participation in the study, those children who

* Have height or weight below the 5th percentile
* Have experienced at least one episode of wheezing when aged 6 months or over
* Have suffered at age 6 months or over, from at least one nocturnal cough episode consisting of 3 (or more) consecutive nights resulting in sleep disturbances in a clinical setting where asthma is likely and other conditions have been excluded
* Have chronic pulmonary diseases of any type, such as, but not limited to, cystic fibrosis, or any cranio-facial abnormality, e.g., cleft palate
* Have a personal history of sleep apnea or who have siblings with a history of sleep apnea
* Are treated with any immunomodulator medication such as, e.g., cyclosporin, cyclophosphamide or FK 506 (Tacrolimus)
* Have received or are receiving allergen - specific immunotherapy
* Suffer from concomitant dermatological disease/condition other than atopic dermatitis, that might interfere with the evaluation of the clinical response for atopic dermatitis
* Have an insufficient wash-out period for the following medications:

  * Intranasal or systemic antihistamines: 3 days,
  * Intranasal or systemic decongestants: 3 days,
  * Loratadine, Desloratadine: 10 days,
  * Chromones: 2 weeks,
  * Oral corticosteroids: 1 month,
  * Chronic use (i.e. cumulatively up to 2 weeks within the last 3 months) of inhaled/intranasal corticosteroids: 1 month,
  * Ketotifen: 1 month,
  * Astemizole: 6 weeks
* Have been treated with any antihistamine, including ketotifen, with daily intake for more than 2 consecutive months in the last 6 months before screening

Subject Exclusion criteria to verify at randomization visit (V2):

• Intake of any prohibited medication listed above during the selection period

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 514 (Actual)
Dates: Start 2002-03-20 (Actual); Primary Completion 2006-03-15 (Actual); Study Completion 2006-03-15 (Actual)

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in March 2002 and concluded in March 2006.
Pre-assignment Details: Participant Flow refers to the Intent-to-treat (ITT) population. 514 subjects were initially randomized, 4 subjects withdrew consent before first study drug intake.
Period: Overall Study
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
Started | 255 | 255
Completed | 215 | 219
Not Completed | 40 | 36
Not completed — Adverse Event | 3 | 6
Not completed — Lost to Follow-up | 8 | 4
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 21 | 22
Not completed — Atopic dermatitis poorly controlled | 0 | 1
Not completed — Eczema deterioration | 0 | 1
Not completed — Parent decision | 1 | 1
Not completed — Investigator decision | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Eczema poorly controlled | 1 | 0
Not completed — Patient relocated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intention-to-Treat (ITT) population.
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Total Title
Number analyzed (Participants) | 255 | 255 | 510
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 255 | 255 | 510
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 19.42 (3.86) | 19.28 (3.94) | 19.35 (3.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 100 | 191
  Male | 164 | 155 | 319

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Asthma During the Treatment Period
Description: The time to onset of asthma was defined as the period elapsed between the randomization visit (V2) and the date of onset of asthma.
  Instead of the median the first Quartile is reported since the median (50%) was not reached.
Time Frame: During the treatment period (18 months)
Population: Intention-to-treat (ITT) population, consisting of all randomized subjects who took at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
Number analyzed (Participants) | 255 | 255
months | NA [9.5 to NA] — Median not reached due to insufficient number of events. | NA [10.3 to NA] — Median not reached due to insufficient number of events.
Statistical Analysis 1: Comparison: Placebo (PBO) vs Levocetirizine (LCTZ); Test type: Superiority or Other; p = 0.991, Regression, Cox; Hazard Ratio (HR) = 1.002, 95% CI 2-sided [0.750 to 1.338]

2. Secondary Outcome: Percentage of Days With Symptoms of Either Wheezing or Nocturnal Cough
Description: The caring person was to note on the diary card each nocturnal cough event with sleep disturbances occurring from 7:00 pm to 7:00 am and each wheezing event occurring at any time together with the treatment for these symptoms.
Time Frame: During the treatment period (18 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
Number analyzed (Participants) | 255 | 255
percentage of days | 3.5 (6.26) | 2.85 (4.53)

3. Secondary Outcome: Percentage of Days With Symptoms of Wheezing
Description: The caring person was to note on the diary card each each wheezing event occurring at any time.
Time Frame: During the treatment period (18 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
Number analyzed (Participants) | 255 | 255
percentage of days | 1.31 (3.00) | 0.88 (1.87)

4. Secondary Outcome: Percentage of Days With Symptoms of Nocturnal Cough
Description: The caring person was to note on the diary card each nocturnal cough event with sleep disturbances occurring from 7:00 pm to 7:00 am
Time Frame: During the treatment period (18 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
Number analyzed (Participants) | 255 | 255
percentage of days | 2.72 (5.24) | 2.33 (4.30)

5. Secondary Outcome: Percentage of Subjects Using Asthma Medication
Description: The following asthma medications were taken into consideration: Beta 2-mimetics, cromoglycates, inhaled corticoids, systemic corticoids, leukotriene antagonists
Time Frame: During the treatment period (18 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
Number analyzed (Participants) | 255 | 255
percentage of participants
  Beta 2 Mimetics | 33.3 | 33.3
  Cromoglycates | 0.8 | 1.2
  Inhaled Corticoids | 18.8 | 15.3
  Systemic Corticoids | 18.4 | 12.5
  Leukotriene antagonists | 2.7 | 3.5

6. Secondary Outcome: Percentage of Days of Use of Asthma Medication
Description: as for outcome 5
Time Frame: During the treatment period (18 months)
Population: 255 subject were included in the Intention-to-treat (ITT) set. Number of participants analyzed is given for each individual category.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
Number analyzed (Participants) | 255 | 255
percentage of days
  Beta 2 Mimetics: number analyzed (Participants) | 249 | 252
  Beta 2 Mimetics | 2.36 (9.31) | 1.37 (4.47)
  Cromoglycates | 0.03 (0.37) | 0.09 (1.24)
  Inhaled Corticoids: number analyzed (Participants) | 252 | 255
  Inhaled Corticoids | 3.60 (12.03) | 1.98 (7.49)
  Systemic Corticoids: number analyzed (Participants) | 254 | 255
  Systemic Corticoids | 0.31 (1.02) | 0.13 (0.45)
  Leukotriene antagonists | 0.30 (2.19) | 0.34 (3.23)

7. Secondary Outcome: Percentage of Subjects Using Medication for Atopic Dermatitis
Description: The following medications for Atopic Dermatitis were taken into consideration: Topical corticosteroids/ Local Steroids Class A, non-steroidal anti-inflammatory (NSAI) creams, tar/ Local Steroids Class B/ Local Steroids Class C/ Topical tacrolimus/ Topical pimecrolimus/ Systemic H1 anti-histamines/ Local antibiotics or antiseptics
Time Frame: During the treatment period (18 months)
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
Number analyzed (Participants) | 255 | 255
percentage of subjects
  Topical corticosteroids | 61.6 | 63.9
  Local Steroids Class A, NSAI creams, tar | 31.4 | 33.3
  Local Steroids Class B | 28.6 | 27.1
  Local Steroids Class C | 33.7 | 37.3
  Topical tacrolimus | 0.8 | 1.2
  Topical pimecrolimus | 2.4 | 5.5
  Systemic H1 anti-histamines | 22.0 | 19.6
  Local antibiotics or antiseptics | 12.9 | 11.0

8. Secondary Outcome: Percentage of Days of Use of Medication for Atopic Dermatitis
Description: The following medications for Atopic Dermatitis were taken into consideration: Emollients, local antihistamines; Local steroids class (LSC) A, non-steroidal anti-inflammatory (NSAI) creams, tar; Local steroids class B; Local steroids class C; Local antibiotics or antiseptics; Oral H1 anti-histamines (a-h); Local antibiotics (ABs) or antiseptics
Time Frame: During the treatment period (18 months)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
Number analyzed (Participants) | 255 | 255
percentage of days
  Topical corticosteroids: number analyzed (Participants) | 223 | 231
  Topical corticosteroids | 32.42 (42.96) | 31.84 (42.70)
  LSC A, NSAI creams, tar: number analyzed (Participants) | 238 | 242
  LSC A, NSAI creams, tar | 15.40 (33.69) | 18.64 (37.30)
  LSC B: number analyzed (Participants) | 240 | 245
  LSC B | 14.23 (32.19) | 12.30 (30.49)
  LSC C: number analyzed (Participants) | 243 | 247
  LSC C | 9.82 (24.98) | 8.27 (22.16)
  Topical tacrolimus: number analyzed (Participants) | 255 | 254
  Topical tacrolimus | 0.36 (5.41) | 0.02 (0.21)
  Topical pimecrolimus: number analyzed (Participants) | 255 | 254
  Topical pimecrolimus | 0.52 (5.62) | 0.31 (2.31)
  Systemic H1 a-h: number analyzed (Participants) | 247 | 252
  Systemic H1 a-h | 3.80 (14.28) | 1.95 (8.84)
  Local ABs or antiseptics: number analyzed (Participants) | 252 | 253
  Local ABs or antiseptics | 2.99 (15.00) | 2.63 (15.37)

9. Secondary Outcome: Percentage of Subjects With Urticaria
Description: Urticaria was defined as typical hives or areas of skin swelling, redness and itching distinctly different from the child's usual inflamed skin lesions of Atopic Dermatitis (AD), associated with an infection or food allergen ingestion/contact or other trigger.
Time Frame: During the treatment period (18 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
Number analyzed (Participants) | 255 | 255
percentage of participants | 41.6 | 27.5

10. Secondary Outcome: Number of Episodes of Urticaria Per Subject
Description: as for outcome 9
Time Frame: During the treatment period (18 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of episodes
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
Number analyzed (Participants) | 255 | 255
Number of episodes | 1.71 (4.05) | 0.71 (1.83)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 1 until during the treatment phase (up to month 18).
Description: Adverse Events refer to the Intention-to-treat (ITT) population, consisting of all randomized subjects who took at least one dose of study medication.
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ)
All-Cause Mortality (participants affected / at risk) | 0/255 | 0/255
Serious Adverse Events (participants affected / at risk) | 37/255 | 31/255
Other Adverse Events (participants affected / at risk) | 240/255 | 239/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PBO) (N=255) | Levocetirizine (LCTZ) (N=255)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1
Bronchitis acute (Infections and infestations) | 0 | 1
Bronchitis chronic (Infections and infestations) | 3 | 0
Bronchopneumonia (Infections and infestations) | 1 | 4
Eczema infected (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 5 | 2
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
Haemophilus infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 19 | 12
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1
Bronchitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PBO) (N=255) | Levocetirizine (LCTZ) (N=255)
Conjunctivitis (Eye disorders) | 41 | 49
Constipation (Gastrointestinal disorders) | 8 | 14
Diarrhoea (Gastrointestinal disorders) | 41 | 48
Teething (Gastrointestinal disorders) | 21 | 22
Vomiting (Gastrointestinal disorders) | 29 | 31
Pyrexia (General disorders) | 71 | 85
Seasonal allergy (Immune system disorders) | 13 | 6
Bronchitis (Infections and infestations) | 52 | 44
Bronchitis acute (Infections and infestations) | 13 | 12
Ear infection (Infections and infestations) | 39 | 38
Gastroenteritis (Infections and infestations) | 55 | 57
Influenza (Infections and infestations) | 18 | 25
Laryngitis (Infections and infestations) | 9 | 19
Nasopharyngitis (Infections and infestations) | 74 | 79
Otitis media (Infections and infestations) | 40 | 36
Pharyngitis (Infections and infestations) | 53 | 58
Respiratory tract infection (Infections and infestations) | 18 | 15
Rhinitis (Infections and infestations) | 71 | 73
Tonsillitis (Infections and infestations) | 28 | 21
Upper respiratory tract infection (Infections and infestations) | 126 | 131
Varicella (Infections and infestations) | 34 | 30
Viral infection (Infections and infestations) | 24 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 67 | 57
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 19 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days